CLINICAL TRIAL: NCT06631248
Title: The Effects of Structured Coordinative Exercise Protocol on Physical Fitness, Motor Competence and Inhibitory Control in Preschool Children
Brief Title: Effects of Coordinative Exercise on Physical Fitness, Motor Competence, and Inhibitory Control in Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, umut canlı, Assoc. Prof., Namik Kemal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NamikemalU
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Motor Skills; Inhibitory Control; Physical Fitness
Keywords: coordination; exercise; preschool children
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The research was divided into groups according to the convenience sampling method. Convenience sampling is a non-random sampling method in which the sample to be selected from the main mass is determined by the judgement of the researcher. In convenience sampling, data are collected from the main mass in the easiest, fastest and most economical way [73,74]. At this point, two classes in the same kindergarten, which accepted to participate in the study and met the conditions for participation in the study, was assigned as the control group (CG; n= 23) and the other class as the exercise group (EG; n= 18).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coordinative exercise protocol (Experimental): coordinative exercise group
  Interventions: Other: Coordinative exercise protocol
- control group (No Intervention): The control group continued the standard education curriculum in kindergarten and did not receive any intervention

INTERVENTIONS:
Other: Coordinative exercise protocol — During the eight-week period, all children in the structured coordinative exercise intervention group participated in 30-minute sessions twice a week on the same day and time. The purpose-oriented basic movement patterns created in the coordinative exercise content were organised in a play-oriented manner suitable for the preschool age range.
  Arms: Coordinative exercise protocol

SUMMARY:
The goal of this study was to determine whether a structured coordinative exercise program could improve physical fitness, motor competence, and inhibitory control in preschool children. The main questions it aimed to answer were:

Does the exercise program improve children's physical fitness (agility, balance, vertical jump)? Does it enhance motor competence, particularly hand-eye coordination and balance? Does it affect inhibitory control, a key component of cognitive function? Researchers compared children who participated in an 8-week exercise program to those who followed their regular school activities.

Participants:

Took part in two 30-minute exercise sessions per week for 8 weeks Were assessed before and after the intervention on physical fitness, motor competence, and inhibitory control The study found significant improvements in physical fitness and motor competence, but no significant changes in inhibitory control.

DETAILED DESCRIPTION:
Scope and Content of the Study

This study evaluated the effectiveness of a structured coordinative exercise protocol aimed at improving physical fitness, motor competence, and inhibitory control in preschool children. Early childhood is considered a critical period for both physical and cognitive development. During this phase, enhancing motor skills and physical fitness forms a crucial foundation for long-term health, social adaptation, and academic success. However, these developmental opportunities may be missed if children do not engage in sufficient levels of physical activity. In this context, the study sought to investigate the effects of exercise interventions that support both motor and cognitive skills in preschool-aged children.

The main goal of the study was to examine how coordinative exercises improve physical fitness and motor competence in preschool children. Additionally, the study explored the impact of these exercises on inhibitory control, a cognitive skill related to attention and impulse control. Inhibitory control is especially important during the preschool years, as it directly affects children's learning processes and social interactions, serving as a key component of executive functions.

Research Protocol and Exercise Intervention

This study was conducted with 41 children, who were randomly assigned to two groups: an exercise group and a control group. The exercise group participated in an 8-week program, consisting of 30-minute sessions twice a week. The program was designed to improve various motor skills such as balance, hand-eye coordination, jumping, and locomotor abilities through play-based activities. The control group continued with their regular school curriculum without additional physical activity interventions.

The exercise protocol included open-ended tasks that progressively moved from simple to complex, requiring movement planning. These play-based exercises aimed to create an engaging and active environment in which children could participate socially. The coordinative exercises focused on supporting a wide range of motor movements and control mechanisms, encouraging the coordination of different body components in harmony.

Assessed Parameters

In the study, children's physical fitness, motor competence, and inhibitory control were assessed both before and after the intervention:

Physical fitness was measured through tests of balance, agility, and vertical jumping.

Motor competence was evaluated using the KTK3+ test battery, which includes tasks such as hand-eye coordination, balancing, and jumping sideways.

Inhibitory control was measured using the Go/No-Go test from the Early Years Toolbox, assessing how well children manage attention and control impulses.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing children
* Participants must not be taking medication
* Must not have any cardiovascular, neurological, orthopaedic or psychiatric disease
* Must be between 5-6 years of age

Exclusion Criteria:

* Having any cardiovascular, neurological, orthopaedic or psychiatric disease
* Having intellectual disability
* Not being between 5-6 years old

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Changes in Motor Competence: KTK3+ Backward Balancing (number of repetitions) | before and at the end of the 8-week intervention.
  Backward balancing is a component of the Körperkoordinationstest für Kinder (KTK3+) motor competence test battery. This test measures the ability to maintain balance while moving backwards on a balance beam.
  Unit of Measurement: number of repetitions (number of backward steps).
Changes in Motor Competence: KTK3+ Move Sideways (Number of repetitions within 20 seconds) | before and at the end of the 8-week intervention.
  Move Sideways, is a component of the Körperkoordinationstest für Kinder (KTK3+) motor competence test battery. This test evaluates the ability to perform coordinated sideways movements.
  Unit of Measurement: Repetitions (Number of repetitions within 20 seconds).
Changes in Motor Competence: KTK3+ Jumping Sideways (Number of repetitions within 15 seconds) | before and at the end of the 8-week intervention.
  jumping sideways is a component of the Körperkoordinationstest für Kinder (KTK3+) motor competence test battery. This test measures the ability to perform coordinated sideways jumps.
  Unit of Measurement: Repetitions (number of repetitions within 15 seconds)
Changes in Motor Competence: KTK3+ Eye-Hand Coordination Task (Number of repetitions within 30 seconds) | before and at the end of the 8-week intervention.
  Eye-Hand Coordination is a component of the Körperkoordinationstest für Kinder (KTK3+) motor competence test battery. This task measures the ability to coordinate visual input with manual responses. It is a measurement method that involves throwing a tennis ball against a wall from a certain distance and holding it with the other hand.
  Unit of Measurement: Number of correct repetitions in 30 seconds.
Changes in Counter Movement Jump Performance, (Highest jump height (cm)) | before and at the end of the 8-week intervention.
  Counter Movement Jump Performance was assessed using an accelerometer system (IVMES Athlete, Ankara, Turkey).
  Unit of Measurement: Centimeter (cm) - Highest jump height
Changes in Balance Performance - Static Balance (%) | before and at the end of the 8-week intervention.
  Balance performance was assessed with a static balance task using a movable platform (Sensbalance MiniBoard; Sensamove®, Utrecht, The Netherlands) that can be connected to a computer.
  Unit of Measurement: Automatically calculated scores in % were used.
Changes in Balance Performance - Dynamic Balance (%) | before and at the end of the 8-week intervention.
  Balance performance was assessed with a dynamic balance task using a moving platform (Sensbalance MiniBoard; Sensamove®, Utrecht, The Netherlands) that can be connected to a computer.
  Unit of Measurement: Automatically calculated scores in % were used.
Changes in Agility (time to complete the test - in seconds) | before and at the end of the 8-week intervention.
  It was evaluated using the Pro-Agility Test. Unit of Measurement: Seconds (s) - Time to complete the test
Changes in Inhibitory Control | before and at the end of the 8-week intervention.
  Inhibitory control was assessed using the Go/No-Go test in the Early Years Toolbox, which measures the ability to suppress inappropriate responses.
  Unit of Measurement: Number of Correct Responses and reaction time of the number of correct responses (ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdag Namik Kemal University, Sports Sciences Research and Development Centre, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the following individual participant data (IPD) from our study:
  Measurements: Data obtained from Physical Fitness, Motor Competence and Inhibitor control parameters will be shared.
  Data Anonymization: All shared IPD will be fully anonymized to protect participant privacy. Personal identifiers such as names, addresses, and contact information will be removed. Data will be aggregated where necessary to prevent re-identification of participants.
  Data Format: The data will be shared in a secure, standardized format (e.g., CSV or Excel files) to facilitate ease of use and analysis by other researchers.
  Access Control: Access to the shared IPD will be granted to qualified researchers who provide a valid research proposal and agree to comply with data use agreements that ensure the data will be used solely for research purposes and not for commercial gain.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Access Control: Access to the shared IPD will be granted to qualified researchers who provide a valid research proposal and agree to comply with data use agreements that ensure the data will be used solely for research purposes and not for commercial gain.

REFERENCES:
- [Background] Chang YK, Tsai YJ, Chen TT, Hung TM. The impacts of coordinative exercise on executive function in kindergarten children: an ERP study. Exp Brain Res. 2013 Mar;225(2):187-96. doi: 10.1007/s00221-012-3360-9. Epub 2012 Dec 13. PMID 23239198
- [Background] Borioni F, Biino V, Tinagli V, Pesce C. Effects of Baby Swimming on Motor and Cognitive Development: A Pilot Trial. Percept Mot Skills. 2022 Aug;129(4):977-1000. doi: 10.1177/00315125221090203. Epub 2022 Apr 26. PMID 35473471
- [Derived] Sendil AM, Canli U, Sheeha BB, Alkhamees NH, Batrakoulis A, Al-Mhanna SB. The effects of structured coordinative exercise protocol on physical fitness, motor competence and inhibitory control in preschool children. Sci Rep. 2024 Nov 18;14(1):28462. doi: 10.1038/s41598-024-79811-3. PMID 39558052